CLINICAL TRIAL: NCT01612962
Title: Diagnostic Tests to Help Determine Osteomyelitis: an Analysis and Comparison of Clinical Signs, Microbiology, Pathology and Radiology.
Brief Title: Diagnostic Tests to Help Determine Osteomyelitis
Status: Terminated | Type: Observational
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, John Steinberg, DPM, Associate Professor, Georgetown University
Other Study IDs: 2011-316
Record Dates: First submitted 2012-05-30; First posted 2012-06-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Osteomyelitis
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bony debridement or amputation: In this study, the investigators will perform a retrospective chart analysis of patients that underwent a bony debridement or amputation in the operating room at Georgetown University Hospital during 2009-2010 under Drs. Steinberg and Attinger

SUMMARY:
In this study, the investigators will perform a retrospective chart analysis of patients that underwent a bony debridement or amputation in the operating room at Georgetown University Hospital during 2009-2010 under Drs. Steinberg and Attinger. Chart reviews, medical records and operative reports via EMR and paper charts will be examined from inpatient records, the Center for Wound Healing, the Emergency Department as well as other institutions involved in the care of the subjects to gather data.

DETAILED DESCRIPTION:
Osteomyelitis is present in approximately 20% of cases of foot infection in persons with diabetes [1, 2] and greatly increases the likelihood that the patient will require a lower-extremity amputation [3, 4]. Early diagnosis and treatment drastically improves prognosis. While there are multiple modalities through which osteomyelitis is diagnosed, unfortunately there is no definitive method. Bone biopsy with histopathological and microbiological analysis has been deemed the gold standard for diagnosing osteomyelitis [3, 5].

Osteomyelitis is considered proven if one or more pathogens are cultured from a reliably obtained bone specimen that shows bone death, acute or chronic inflammation and reparative responses on histological examination. However, histological analysis can also produce falsely positive results based on sampling error or if there are other causes of inflammation [6]. Furthermore, a recent study done by Meyr et al. has highlighted a discrepancy amongst pathologists that leaves the medical community questioning the validity of some pathological diagnoses.

Microbiological analysis can differ based on specimen processing and is also dependent on sampling technique. Often results can be falsely negative because of sampling error, prior antibiotic therapy, or inability to culture fastidious organisms; likewise, they may be falsely positive because of contamination by wound-colonizing flora [6].

Also, cultures of superficial swab samples from diabetic ulcers and sinus tracts may not adequately identify the true bacteriological characteristics of diabetic foot osteomyelitis because of bacterial colonization of the wound surfaces with microorganisms that are typically not considered to be pathogenic (such as enterococci and coagulase-negative staphylococci) [7]. Senneville et al. attempted to define the true correlation between cultures of swab samples and cultures of bone biopsy specimens obtained from areas of osteomyelitis in the diabetic foot. It was found that swab cultures are inaccurate and unreliable indicators of the pathogenic organism in chronic diabetic foot osteomyelitis and there was overall poor concordance between the superficial swab culture and bone biopsy culture results for all microorganisms [8].

Other methods for diagnosing osteomyelitis include radiographic analysis. On plain film, osteomyelitis is suspected when one or more of the following radiographic signs is observed: periosteal elevation, cortical disruption, medullary involvement, osteolysis, and sequestra (segments of necrotic bone separated from living bone by granulation tissue) [9]. Signs of osteomyelitis only show up on plain film 10-20 days after infection, [10, 11]. Dinh et al, in their meta-analysis on radiographic modalities, found 54% sensitivity and 68% specificity in detecting osteomyelitis with plain film versus 90% sensitivity and 79% specificity with MRI [12].

To the investigators' knowledge, there has been no study that compares all these methods to determine if there is a superior test to determine osteomyelitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients that underwent a bony debridement or amputation in the operating room at Georgetown University Hospital during 2009-2010 under Drs. Steinberg and Attinger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that underwent a bony debridement or amputation in the operating room at Georgetown University Hospital during 2009-2010 under Drs. Steinberg and Attinger
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2011-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Accuracy of Osteomyelitis Diagnostic Testing | 12 months
  The purpose of this study is to help compare accuracy of all the diagnostic tests that are used in current practice to help determine osteomyelitis.

SECONDARY OUTCOMES:
Reliability of diagnostic testing for Osteomyelitis | 12 months
  To find a test that is the most reliable in determining osteomyelitis

CONTACTS AND LOCATIONS:
Overall Officials: John J. Steinberg, DPM, Principal Investigator — Georgetown University Hospital; Paul Kim, DPM, Study Director — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States